CLINICAL TRIAL: NCT02683486
Title: The Assessment of Intelligent Oxygen Therapy (iO2T) in Patients on Long-term Oxygen Therapy During Activities of Daily Living
Brief Title: Intelligent Oxygen Therapy During Activities of Daily Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 15IC2835
Record Dates: First submitted 2016-01-26; First posted 2016-02-17 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Hypoxia; COPD; Hyperoxia
MeSH Terms: conditions — Hypoxia; Pulmonary Disease, Chronic Obstructive; Hyperoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Activities of daily living on iO2t (Experimental): Patients will complete simulated activities of daily living on intelligent oxygen therapy (an auto-titrating oxygen system)
  Interventions: Device: Intelligent oxygen therapy (an auto-titrating oxygen system)
- Activities of daily living on LTOT (Active Comparator): Patients will complete activities of daily living on their usual long-term oxygen therapy.
  Interventions: Device: Long-term oxygen therapy

INTERVENTIONS:
Device: Intelligent oxygen therapy (an auto-titrating oxygen system) — This device is an auto-titrating oxygen system. The system is programmed to maintain a specific target SpO2 by automatically adjusting the oxygen flow rate. The system can deliver flow rates of 0-5 litres/minute.
  Arms: Activities of daily living on iO2t
Device: Long-term oxygen therapy — This is the patients usual long-term oxygen therapy
  Arms: Activities of daily living on LTOT

SUMMARY:
The aim of this study is to assess whether an auto-titrating oxygen system can maintain constant oxygen saturations (SpO2) in patients who are on long-term oxygen therapy (LTOT) during activities of daily living.

Currently LTOT is provided at a constant fixed-flow rate e.g. 2 litres per minute all the time after appropriate assessment. The flow rate is not changed during usual household activities but is increased for walking. A number of studies have investigated the SpO2 of patients on LTOT during the daytime in patients' homes. The results have shown that patients' SpO2 decreases intermittently whilst they are doing activities of daily living such as watching television, putting away the shopping, having a shower or bath and dressing and undressing. This is a problem as it can lead to breathlessness, increased stress on the heart and affect brain function. In order to correct the drop in SpO2 that patients experience during everyday activities, the investigators have developed an oxygen system, which can automatically change the amount of oxygen delivered depending on a patients' oxygen saturations - an auto-titrating oxygen system. In this study, patients on LTOT will be asked to simulate a series of activities of daily living twice: once whilst on their usual fixed-flow oxygen therapy and once on the auto-titrating oxygen system. The activities will be carried out in a hospital setting. During the activities, SpO2 will be recorded continuously. The main outcome of interest from the study will be the SpO2 throughout the study on fixed-flow oxygen and the auto-titrating oxygen system.

DETAILED DESCRIPTION:
Long-term oxygen therapy (LTOT) is prescribed for patients with stable severe hypoxemic respiratory failure according to specific criteria set out in different guidelines from international respiratory societies. The aim of LTOT is to maintain the resting partial pressure of oxygen (PO2) >60 mmHg or oxygen saturation (SpO2) >90%.

A number of studies have demonstrated that whilst at home, patients on LTOT experience episodes of intermittent hypoxia (SpO2 <90%) and spend significant amounts of time with SpO2 <90%. These episodes of desaturation occur most frequently during activities of daily living and may be harmful as they could lead to pulmonary hypertension, arrhythmias and ischaemic heart disease. Simply increasing the LTOT flow rate by 1 or 2 litres in one option but this exposed the patients to hyperoxaemia and the risk of hypercapnia. An another method optimising LTOT is to utilise an auto-titrating oxygen system. These system allow close control of SpO2 by automatically adjusting the flow of oxygen to match a target SpO2. At the Royal Brompton Hospital and Imperial College London, the investigators have developed our own auto-titrating oxygen system - called intelligent oxygen therapy (iO2t).

This system has been tested in patients with chronic obstructive pulmonary disease (COPD) and LTOT during a 6 minute walk test with promising results (ERS 2015).

The aim of this study is to investigate whether the intelligent oxygen therapy system can reduce intermittent hypoxia in patients on LTOT during simulated activities of daily living. Patients will be asked to a series of activities of daily living over a period of 1 hour including: washing, dressing, putting away shopping and cleaning. The patients will do these activities twice: once on their usual LTOT and once on the auto-titrating oxygen system in a cross-over design.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Currently on or eligible for LTOT for respiratory failure

Exclusion Criteria:

1. LTOT flow rate ≥4 litres per minute
2. Exacerbation of underlying lung disease in the past 4 weeks
3. Inability to understand English
4. Significant co-morbidities
5. Patients who lack capacity to consent
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
The percentage of time spent with SpO2 <90% during the activities of daily living - 55 minutes | Calculated over the duration of the time the patient is carrying out activities of daily living (55 minutes)

SECONDARY OUTCOMES:
Mean SpO2 during the activities of daily living - 55 minutes | Calculated over the duration of the time the patient is carrying out activities of daily living (55 minutes)
Mean Heart rate during the activities of daily living - 55 minutes | Calculated over the duration of the time the patient is carrying out activities of daily living (55 minutes)
Borg score for breathlessness and fatigue at the end of activities of daily living (55 minutes) | At the end of activities of daily living (55 minutes)
Total volume of oxygen delivered during simulated activities of daily living during the activities of daily living (55 minutes) | Calculated over the duration of the time the patient is carrying out activities of daily living (55 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Simonds, FRCP, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton and Harefield NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mohammad Moghal, Rishi Goburdhun, Mary Morrell, Robert Dickinson, Anita Simonds A Novel Smartphone Based Auto-Titrating Oxygen System Reduces Intermittent Hypoxia During Activities of Daily Living in Patients on Long-Term Oxygen Therapy. American Journal of Respiratory and Critical Care Medicine 2017;195:A7709
- See also: This is link to PhD thesis of M Moghal showing results of study on Intelligent Oxygen therapy during Activities of Daily Living — https://spiral.imperial.ac.uk/handle/10044/1/59707